CLINICAL TRIAL: NCT07103967
Title: Investigating the Effect of Alcohol Serving Size and Calorie Information on Alcohol Consumption: A Real-world Experiment
Brief Title: Investigating the Effects of Calorie Information and Serving Size of Alcohol Products on Alcohol Consumption.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liverpool (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AlcCal Real-world Study
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-07

CONDITIONS: Obesity and Overweight; Alcohol
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Calorie information present, serving size reduced (Experimental): Participants will be presented with calorie information of alcohol products, and will have a restricted selection of serving sizes of drinks available to them.
  Interventions: Behavioral: Calorie information manipulation; Behavioral: Serving size manipulation
- Calorie information present, serving size typical (Experimental): Participants will be presented with calorie information of alcohol products, and the serving sizes of drinks available to participants will not be manipulated.
  Interventions: Behavioral: Calorie information manipulation; Behavioral: Serving size manipulation
- Calorie information absent, serving size reduced (Experimental): Participants will not be presented with calorie information of alcohol products, and will have a restricted selection of serving sizes of drinks available to them.
  Interventions: Behavioral: Calorie information manipulation; Behavioral: Serving size manipulation
- Calorie information absent, serving size typical (Experimental): Participants will not be presented with calorie information of alcohol products, and the serving sizes of drinks available to participants will not be manipulated.
  Interventions: Behavioral: Calorie information manipulation; Behavioral: Serving size manipulation

INTERVENTIONS:
Behavioral: Calorie information manipulation — The intervention will be administered by changing the information presenting to participants at point-of-choice when ordering alcoholic drinks and bar snacks. When alcohol calorie information is present, participants will see the calorie content of alcohol products on menus and at other point-of-choice locations. When it is not present, this information will be absent.
Behavioral: Serving size manipulation — The intervention will be administered by changing the availability of alcoholic drinks. When serving sizes are reduced, participants will only be able to order 2/3 pint of 1/2 servings of beer, and 125 ml servings of wine. When serving sizes are not reduced, participants will be able to order 1 pint servings or 1/2 servings of beer, and 175 ml or 125 ml servings of wine.

SUMMARY:
The present study aims to investigate whether alcohol consumption is reduced when participants are shown calorie information of alcohol products, compared with when calorie information is absent. We also wish to see whether alcohol consumption levels are reduced when changing the serving sizes available to participants.

DETAILED DESCRIPTION:
We will examine the effect of alcohol calorie information on calorie and alcohol unit consumption in a semi-naturalistic real-world experiment by randomising pub quiz evenings to alcohol calorie information vs. absence of calorie information (control). Because current evidence for alcohol calorie information from online hypothetical choice experiments suggests any impact on alcohol consumption may be null or very small, we will compare and benchmark the size of any potential effect of alcohol calorie information to another public health alcohol intervention known to reduce alcohol consumption (alcohol serving size). We will achieve this by also randomizing evenings to normal sized servings of alcohol (control) vs. reduced serving sizes. In addition to examining effects of interventions on what people drink and eat during the pub quiz, we will examine alcohol and energy intake after the pub quiz to probe for potential compensatory behaviour in response to interventions. Because it is currently unclear how useful consumers find alcohol information when implemented in real-world conditions, we will also examine the extent to which participants perceive the interventions to be effective.

ELIGIBILITY:
Inclusion Criteria:

* Consume alcohol on a regular basis (at least one UK unit per week)
* Be aged 18 or over

Exclusion Criteria:

* Have a current or previously diagnosed alcohol use disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2025-11-19 (Estimated); Study Completion 2025-11-19 (Estimated)

PRIMARY OUTCOMES:
Alcohol units | Duration of the evening (approximately 3 hours and 15 minutes)
  Amount of alcohol units consumed in the evening.
Total calorie consumption | Duration of the evening (approximately 3 hours and 15 minutes)
  The amount of calories consumed during the evening.

SECONDARY OUTCOMES:
Perceived message effectiveness | The day after the intervention
  Participants will be asked to rate whether the menu they were presented with, affected feelings of concern towards alcohol.
Follow-up energy intake | Immediately after the intervention
  Participants will be asked to record the food and drink consumed immediately after leaving the pub quiz, for the rest of the evening.
Bar snack consumption (calories) | Duration of the evening (approximately 3 hours and 15 minutes)
  The amount of snacks consumed during the evening will be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Liverpool, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
An anonymised data set will be published on the open science framework for anyone to access.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be available after data collection has finished, this will be available indefinitely.